CLINICAL TRIAL: NCT02437760
Title: Determination of the Prognostic and Predictive Value of the Cancer Antigen-125 (CA-125) Marker in Lung Cancer Monitoring
Brief Title: The Prognostic and Predictive Value of the CA-125 Marker in Lung Cancer Monitoring
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: E-DA Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EMRP49103N
Record Dates: First submitted 2015-04-18; First posted 2015-05-08 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: serum and pleural effusion CA-125 level — serum and pleural effusion(if exist) CA-125 are collected:
  * at time of diagnosis
  * every 3 month during treatment
  * stop at the progression or after 12 months

SUMMARY:
The tumor associated CA-125antigen for diagnosis and follow-up of ovarian cancer was well defined. Increased serum CA125 level may have many diagnoses other than ovarian cancer, including breast, colorectal and lung cancer. 80% lung cancer patients were diagnosed at advanced stage. Malignant pleural effusion secondary to lung cancer represented the condition of cancer cell involved pleura.

The CA-125 level may reflect the extent of tumor involved in pleura (tumor burden), it could be correlated with the prognosis. This study was performed to examine the properties of CA-125 by measuring pleural and blood CA-125 levels in lung cancer with or without malignant pleural effusion; meanwhile to examine whether the rate of decline in CA 125 during primary therapy as a surrogate indicator for survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proved lung cancer

Exclusion Criteria:

* History of other cancers within the past 5 years
* Pregnancy or breast milk feeding
* TB pleuritis and peritonitis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with histologically proved lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
The diagnostic Value of the cancer antigen-125 in lung cancer | 12months
  1. Comparison of CA-125 level in serum between lung cancer patients with or without malignant pleural effusion
  2. The correlation between serum and pleural effusion CA-125 level

SECONDARY OUTCOMES:
The prognostic value of the cancer antigen-125 in lung cancer | 24 months
  1. Association of serum/ pleural effusion CA-125 level with Disease-Free Survival and Overall Survival
  2. The correlation of CA-125 response at the 3rd , the 6th month between tumor lesion change
  3. Analysis of survival in relation to CA-125 response

CONTACTS AND LOCATIONS:
Locations (1):
- E-DA hospital, Kaohsiung City, Taiwan